CLINICAL TRIAL: NCT00543998
Title: Near Infrared Transillumination of the Paranasal Sinuses
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, B.J Wong, M.D.,Ph.D., Professor Department of Otolaryngology, University of California, Irvine
Other Study IDs: 20022672
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sinusitis
Keywords: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optical Measurement transillumination: Optical Measurement of sinus
  Interventions: Device: Optical Measurement transillumination

INTERVENTIONS:
Device: Optical Measurement transillumination — Optical Measurement of sinus

SUMMARY:
This research project designed to diagnose sinusitis using a simple and low-cost optical tool. Healthy sinuses are typically filled with air, and show up as bright spots on the camera. Infected sinuses are filled with fluid and show up dark spots on the camera. Images of infected sinuses could be used to diagnose sinusitis, or to check if surgical treatments on the sinuses have been successful.

DETAILED DESCRIPTION:
This device consists of a specialized flashlight that uses mostly non-visible light, and a small camera to record the light. The tool is the size and shape of spoon. The technique of shining light into the mouth, face, and sinuses is known as "transillumination" and has been used for nearly a century to aid in the diagnosis of sinusitis. The tool described in this study is a custom made device that uses light that is invisible to the eye.

ELIGIBILITY:
Inclusion Criteria:

* male and female age of 15 years or older.
* Has diagnose of sinusitis, nasal allergies,nasal breathing problem, and tumors.

Exclusion Criteria:

* Age less than 15 year sold

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic,
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2003-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Healthy Sinus | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian JF Wong, M.D.,Ph.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (2):
- United States (2):
  - Beckman Laser Institute Medical Cinic, University of California,Irvine, Irvine, California
  - Otolaryngology Medical Clinic, University of California, Irvine, Irvine, California